CLINICAL TRIAL: NCT05812157
Title: Optimization of Anti-IL17 Antibody Therapy by Associating Fiber Supplementation to Correct Treatment-aggravated Gut Dysbiosis in Axial Spondyloarthritis - RESPOND-IL17
Brief Title: Optimizing Anti-IL17 Antibody Therapy by Associating Fiber Supplementation to Correct Treatment-aggravated Gut Dysbiosis in Axial Spondyloarthritis - RESPOND-IL17
Acronym: RESPOND-IL17
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDRCB : 2022-A00135-38
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Axial Spondyloarthritis
Keywords: dysbiosis; short-chain fatty acids; fiber; microbiota
MeSH Terms: conditions — Axial Spondyloarthritis; Dysbiosis

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, prospective, randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All treatments will be numbered. The treatment number will be assigned according to the randomization list. All participants (patient/evaluator/etc.) will be blinded to the treatment administered. Only the hospital pharmacy will know the assigned treatment and will guarantee the blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients with aSp receiving fiber supplements in the form of Fibruline® Instant (Fagron laboratories)
  Interventions: Dietary Supplement: Daily dietary supplementation with Fibruline; Drug: Anti-IL-17 therapy
- Control group (Placebo Comparator): Patients with aSp receiving fake fiber supplements (placebo) in the form of Maltodextrine (laboratoire Fagron).
  Interventions: Dietary Supplement: Daily dietary supplementation with Fibruline; Drug: Anti-IL-17 therapy

INTERVENTIONS:
Dietary Supplement: Daily dietary supplementation with Fibruline — Supplementation with 12 grams per day of Fibruline reconstituted with 60mL of water, once a day
Drug: Anti-IL-17 therapy — Patients in both groups will be on anti-IL-17 therapy

SUMMARY:
Fiber is the main source of energy for colonic bacteria and its consumption favorably modifies the composition of the microbiota in only a few days. Their fermentation in the colon releases short-chain fatty acids (SCFAs). Clostridiales contain many strains producing SCFAs. These SCFAs can restore the intestinal barrier and promote certain anti-inflammatory cells, including regulatory T cells (Tregs), which are essential to the mechanisms in tolerance of the self. Fibers could therefore correct the intestinal abnormalities present in patients with axial spondyloarthritis (AxSpA) and aggravated by anti-IL-17 drugs and thus improve the therapeutic response to these treatments.

The hypothesis is that dietary fiber will correct the dysbiosis in AxSpA patients and increase the release of SCFAs, which favorably modulate the immune response and improve AxSpA.

DETAILED DESCRIPTION:
Axial spondyloarthritis (AxSpA) is the second most common chronic inflammatory rheumatic disease, which develops preferentially in young subjects and results in a significant impairment of quality of life, particularly due to painful symptoms. The importance of the digestive system has long been recognized, since this disease is considered to be part of a larger group of diseases including Crohn's disease and ulcerative colitis because of their frequent association in the same patient, and because leaky gut disorders and alterations of the intestinal microbiota (dysbiosis) have been described in these patients. These abnormalities may stimulate the immune system and therefore be involved in inflammatory processes (especially Th17). The available treatments are based on non-steroidal anti-inflammatory drugs, and in the event of failure or intolerance, biomedicines targeting TNF can be used. Therapeutic monoclonal antibodies against IL-17 have recently enriched the therapeutic arsenal. Although most anti-TNF agents have a beneficial effect on the rheumatologic and digestive aspects of these diseases, anti-IL-17 agents are not expected to be effective in inflammatory bowel diseases.

Indeed, a deleterious role of anti-IL-17 on the intestinal microbiota has even been demonstrated, which could result in a reduction of the systemic anti-inflammatory effect expected from these molecules, and consequently of the clinical benefit felt by the patient. In fact, anti-IL-17s lead to a significant decrease in Clostridiales, bacteria that participate in intestinal homeostasis.

Fiber is the main source of energy for colonic bacteria and its consumption favorably modifies the composition of the microbiota in just a few days. Their fermentation in the colon releases short-chain fatty acids (SCFAs). Clostridiales contain many strains producing SCFAs. These SCFAs can restore the intestinal barrier and promote certain anti-inflammatory cells, including regulatory T cells (Tregs), which are essential to the mechanisms in tolerance of the self. Fibers could therefore correct the intestinal abnormalities present in AxSpA patients and aggravated by anti-IL-17 drugs and thus improve the therapeutic response to these treatments.

The hypothesis is therefore that dietary fiber will correct the dysbiosis in AxSpA patients and increase the release of SCFAs, which favorably modulate the immune response and thus improve AxSpA.

ELIGIBILITY:
Inclusion criteria:

* Patients with spondyloarthritis meeting the ASAS criteria
* Patient considered by the treating rheumatologist for anti-IL-17 biomedication
* Patients aged between 18 and 90 years of age
* Patients who are affiliated to a French social security system or beneficiaries of such a system
* Patients with no desire to become pregnant during the study period (Effective contraception for women of childbearing age during the study period (surgical sterilization, hormonal contraceptives, barrier method, intrauterine device))

Exclusion Criteria:

* Lack of written informed consent after a time of reflection
* Patients participating in other therapeutic research or having participated in research for which the exclusion period has not ended
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Pregnant or breastfeeding woman
* Patients with digestive disorders for which a chronic inflammatory bowel disease has not been excluded
* Patients with fructose intolerance or glucose or galactose malabsorption
* Patients with known intolerance to inulin or maltodextrin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Clostridial changes in the Experimental group | Week 0
  Patients will receive fiber supplementation with inulin (Fibruline® Instant, Fagron laboratory) at a rate of 12 grams of powder per day reconstituted with approximately 60mL of water and consumed in one intake per day. To confirm the efficacy of treatment, the percentage of patients with a >10% decrease in Clostriadiales in their stools at 3 months after initiation of anti-IL-17 will be recorded. This percentage will be based on the distribution of bacteria analyzed by 16S RNA sequencing.
Clostridial changes in Controls | Week 0
  Patients will receive a placebo consisting of Maltodextrin (Fagron laboratories), packaged in jars identical to those used for inulin, with a volumetric equivalent, an energy contribution and very similar color. Patients will consume 12 grams of powder per day reconstituted with approximately 60mL of water and consumed in one intake per day. The percentage of patients with a >10% decrease in Clostriadiales in their stools at 3 months after initiation of anti-IL-17 will be recorded. This percentage will be based on the distribution of bacteria analyzed by 16S RNA sequencing.
Clostridial changes in the Experimental group | Week 12
  Patients will receive fiber supplementation with inulin (Fibruline® Instant, Fagron laboratory) at a rate of 12 grams of powder per day reconstituted with approximately 60mL of water and consumed in one intake per day. To confirm the efficacy of treatment, the percentage of patients with a >10% decrease in Clostriadiales in their stools at 3 months after initiation of anti-IL-17 will be recorded. This percentage will be based on the distribution of bacteria analyzed by 16S RNA sequencing.
Clostridial changes in Controls | Week 12
  Patients will receive a placebo consisting of Maltodextrin (Fagron laboratories), packaged in jars identical to those used for inulin, with a volumetric equivalent, an energy contribution and very similar color. Patients will consume 12 grams of powder per day reconstituted with approximately 60mL of water and consumed in one intake per day. The percentage of patients with a >10% decrease in Clostriadiales in their stools at 3 months after initiation of anti-IL-17 will be recorded. This percentage will be based on the distribution of bacteria analyzed by 16S RNA sequencing.

SECONDARY OUTCOMES:
Effect of fiber supplementation on clinical therapeutic response in the experimental group: Delta BASDAI | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) will be used to measure the percentage of patients responding positively to treatment.
Effect of fiber supplementation on clinical therapeutic response in the experimental group: Delta BASDAI | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) will be used to measure the percentage of patients responding positively to treatment.
Effect of fiber supplementation on clinical therapeutic response in the experimental group: ASAS20 | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The ASAS20 will be used to measure the percentage of patients responding positively to treatment. This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 20) is defined as an improvement in at least 20% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect of fiber supplementation on clinical therapeutic response in the experimental group: ASAS20 | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The ASAS20 will be used to measure the percentage of patients responding positively to treatment. This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 20) is defined as an improvement in at least 20% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect of fiber supplementation on clinical therapeutic response in the experimental group: ASAS40 | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The ASAS40 will be used to measure the percentage of patients responding positively to treatment. This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 40) is defined as an improvement in at least 40% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect of fiber supplementation on clinical therapeutic response in the experimental group: ASAS40 | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The ASAS40 will be used to measure the percentage of patients responding positively to treatment. This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 40) is defined as an improvement in at least 40% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect of fiber supplementation on clinical therapeutic response in the experimental group: ASDAS | Week 0
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The ASDAS (Ankylosing Spondylitis Disease Activity Score) will be used to measure the percentage of patients responding positively to treatment. This tool is an index to assess disease activity in Ankylosing Spondylitis. The preferred score uses CRP (C-reactive protein) rather than ESR (erythrocyte sedimentation rate).
Effect of fiber supplementation on clinical therapeutic response in the experimental group: ASDAS | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  The ASDAS (Ankylosing Spondylitis Disease Activity Score) will be used to measure the percentage of patients responding positively to treatment. This tool is an index to assess disease activity in Ankylosing Spondylitis. The preferred score uses CRP (C-reactive protein) rather than ESR (erythrocyte sedimentation rate).
Effect of fiber supplementation on clinical therapeutic response: GIQLI | Week 0
  Clinical response rates in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  Digestive symptoms will be assessed using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire at Week 0 and Week 12. The GIQLI is a measure of the subjective perception of well-being by a patient, which may vary unexpectedly between diagnostic groups. The GIQLI was initiated in Germany and includes 36 items asking about symptoms, physical status, emotions, social dysfunction, and effects of medical treatment. The Questions cover the following 5 dimensions : symptoms, physical condition, emotions, social integration and medical treatment.
Effect of fiber supplmentation on clinical therapeutic response: GIQLI | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 with fiber supplementation will be recorded as a percentage.
  Digestive symptoms will be assessed using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire at Week 0 and Week 12. The GIQLI is a measure of the subjective perception of well-being by a patient, which may vary unexpectedly between diagnostic groups. The GIQLI was initiated in Germany and includes 36 items asking about symptoms, physical status, emotions, social dysfunction, and effects of medical treatment. The Questions cover the following 5 dimensions : symptoms, physical condition, emotions, social integration and medical treatment.
Effect at 12 weeks of placebo on clinical therapeutic response: Delta BASDAI | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) will be used to measure the percentage of patients responding positively to treatment.
Effect at 12 weeks of placebo on clinical therapeutic response: Delta BASDAI | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) will be used to measure the percentage of patients responding positively to treatment.
Effect at 12 weeks of placebo on clinical therapeutic response: ASA20 | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  The ASAS20 will be used to measure the percentage of patients responding positively to treatment.This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 20) is defined as an improvement in at least 20% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect at 12 weeks of placebo on clinical therapeutic response: ASA20 | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  The ASAS20 will be used to measure the percentage of patients responding positively to treatment.This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 20) is defined as an improvement in at least 20% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect at 12 weeks of placebo on clinical therapeutic response: ASA40 | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  The ASAS40 will be used to measure the percentage of patients responding positively to treatment.This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 40) is defined as an improvement in at least 40% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect at 12 weeks of placebo on clinical therapeutic response: ASA40 | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  The ASAS40 will be used to measure the percentage of patients responding positively to treatment.This tool was developed by the Assessment of SpondylArthritis international Society (ASAS). The ASAS Response Criteria (ASAS 40) is defined as an improvement in at least 40% and an absolute improvement in at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation (last 2 questions of BASDAI).
Effect at 12 weeks of placebo on clinical therapeutic response: ASDAS | Week 0
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage. The ASDAS (Ankylosing Spondylitis Disease Activity Score) will be used to measure the percentage of patients responding positively to treatment. This tool is an index to assess disease activity in Ankylosing Spondylitis. The preferred score uses CRP (C-reactive protein) rather than ESR (erythrocyte sedimentation rate).
Effect at 12 weeks of placebo on clinical therapeutic response: ASDAS | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage. The ASDAS (Ankylosing Spondylitis Disease Activity Score) will be used to measure the percentage of patients responding positively to treatment. This tool is an index to assess disease activity in Ankylosing Spondylitis. The preferred score uses CRP (C-reactive protein) rather than ESR (erythrocyte sedimentation rate).
Effect of placebo on clinical therapeutic response: GIQLI | Week 0
  Clinical response rates observed in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  Digestive symptoms will be assessed using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire at Week 0 and Week 12. The GIQLI is a measure of the subjective perception of well-being by a patient, which may vary unexpectedly between diagnostic groups. The GIQLI was initiated in Germany and includes 36 items asking about symptoms, physical status, emotions, social dysfunction, and effects of medical treatment. The Questions cover the following 5 dimensions : symptoms, physical condition, emotions, social integration and medical treatment.
Effect of placebo on clinical therapeutic response: GIQLI | Week 12
  Clinical response rates observed at 3 months in patients treated with anti-IL-17 without fiber supplementation will be recorded as a percentage.
  Digestive symptoms will be assessed using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire at Week 0 and Week 12. The GIQLI is a measure of the subjective perception of well-being by a patient, which may vary unexpectedly between diagnostic groups. The GIQLI was initiated in Germany and includes 36 items asking about symptoms, physical status, emotions, social dysfunction, and effects of medical treatment. The Questions cover the following 5 dimensions : symptoms, physical condition, emotions, social integration and medical treatment.
Tolerance of anti-IL17 intervention and treatment in the experimental group: Permeability | Month 0
  Changes in serum concentrations of intestinal permeability markers (zonulin, claudin-3, iFABP); and endotoxemia (LBP, CD14s) will be measured by ELISA in ng/ml
Tolerance of anti-IL17 intervention and treatment in controls: Permeability | Month 3
  Changes in serum concentrations of intestinal permeability markers (zonulin, claudin-3, iFABP); and endotoxemia (LBP, CD14s) will be measured by ELISA in ng/ml
Tolerance of anti-IL17 intervention and treatment in the experimental group | Month 3
  The distribution and diversity of different germs will be measured by 16S RNA sequencing.
  Quantitative
Tolerance of anti-IL17 intervention and treatment in controls | Month 3
  The distribution and diversity of different germs will be measured by 16S RNA sequencing.
  Quantitative
Presence of candida in patients in the experimental group | Month 3
  YES/NO
Presence of candida in patients in the control group | Month 3
  YES/NO
Tolerance of treatment in the experimental group | Month 3
  All adverse events related or not to anti-IL17 treatment and potentially associated with the consumption of high doses of fiber (bloating, flatulence, diarrhea, abdominal pain) will be recorded
Tolerance of treatment in the control group | Month 3
  All adverse events related or not to anti-IL17 treatment and potentially associated with the consumption of high doses of fiber (bloating, flatulence, diarrhea, abdominal pain) will be recorded
Complete blood count: Red blood cells in the experimental group | Month 0
  Red blood cells will be measured in millions/mm3
Complete blood count: Red blood cells in the control group | Month 0
  Red blood cells will be measured in millions/mm3
Complete blood count: Red blood cells in the experimental group | Month 3
  Red blood cells will be measured in millions/mm3
Complete blood count: Red blood cells in the control group | Month 3
  Red blood cells will be measured in millions/mm3
Complete blood count: White blood cells in the experimental group | Month 0
  White blood cells will be measured in millions/mm3
Complete blood count: White blood cells in the control group | Month 0
  White blood cells will be measured in millions/mm3
Complete blood count: White blood cells in the experimental group | Month 3
  White blood cells will be measured in millions/mm3
Complete blood count: White blood cells in the control group | Month 3
  White blood cells will be measured in millions/mm3
Complete blood count: Hemoglobin in the experimental group | Month 0
  Hemoglobin will be measured in g/L
Complete blood count: Hemoglobin in the control group | Month 0
  Hemoglobin will be measured in g/L
Complete blood count: Hemoglobin in the experimental group | Month 3
  Hemoglobin will be measured in g/L
Complete blood count: Hemoglobin in the control group | Month 3
  Hemoglobin will be measured in g/L
Complete blood count: Hematocrit in the experimental group | Month 0
  Hematocrit will be measured as a % of whole blood
Complete blood count: Hematocrit in the control group | Month 0
  Hematocrit will be measured as a % of whole blood
Complete blood count: Hematocrit in the experimental group | Month 3
  Hematocrit will be measured as a % of whole blood
Complete blood count: Hematocrit in the control group | Month 3
  Hematocrit will be measured as a % of whole blood
Complete blood count: Platelets in the experimental group | Month 0
  Platelets will be measured in K/µL
Complete blood count: Platelets in the control group | Month 0
  Platelets will be measured in K/µL
Complete blood count: Platelets in the experimental group | Month 3
  Platelets will be measured in K/µL
Complete blood count: Platelets in the control group | Month 3
  Platelets will be measured in K/µL
T-lymphocytes in the experimental group | Month 0
  The phenotype of T-lymphocytes (Treg, Thelpers) will be measured as % of total white blood cells
T-lymphocytes in the control group | Month 0
  The phenotype of T-lymphocytes (Treg, Thelpers) will be measured as % of total white blood cells
T-lymphocytes in the experimental group | Month 3
  The phenotype of T-lymphocytes (Treg, Thelpers) will be measured as % of total white blood cells
T-lymphocytes in the control group | Month 3
  The phenotype of T-lymphocytes (Treg, Thelpers) will be measured as % of total white blood cells
Monocytes in the experimental group | Month 0
  Monocytes will be measured by flow cytometry (CD25, CD127, CXCR3, CCR6, CD294, CD14, CD16, TNF, IL-6) as % of total white blood cells
Monocytes in the control group | Month 0
  Monocytes will be measured by flow cytometry (CD25, CD127, CXCR3, CCR6, CD294, CD14, CD16, TNF, IL-6) as % of total white blood cells
Monocytes in the experimental group | Month 3
  Monocytes will be measured by flow cytometry (CD25, CD127, CXCR3, CCR6, CD294, CD14, CD16, TNF, IL-6) as % of total white blood cells
Monocytes in the control group | Month 3
  Monocytes will be measured by flow cytometry (CD25, CD127, CXCR3, CCR6, CD294, CD14, CD16, TNF, IL-6) as % of total white blood cells
Aspartate aminotransferase (ASAT) in the experimental group | Month 0
  Aspartate aminotransferase (or ASAT) will be measured in international units per liter
Aspartate aminotransferase (ASAT) in the experimental group | Month 3
  Aspartate aminotransferase (or ASAT) will be measured in international units per liter
Aspartate aminotransferase (ASAT) in the control group | Month 0
  Aspartate aminotransferase (or ASAT) will be measured in international units per liter
Aspartate aminotransferase (ASAT) in the control group | Month 3
  Aspartate aminotransferase (or ASAT) will be measured in international units per liter
Alanine aminotransferase (ALAT) in the experimental group | Month 0
  Alanine aminotransferase (ALAT) will be measured in international units per liter
Alanine aminotransferase (ALAT) in the experimental group | Month 3
  Alanine aminotransferase (ALAT) will be measured in international units per liter
Alanine aminotransferase (ALAT) in the control group | Month 0
  Alanine aminotransferase (ALAT) will be measured in international units per liter
Alanine aminotransferase (ALAT) in the control group | Month 3
  Alanine aminotransferase (ALAT) will be measured in international units per liter
Alkaline phosphatase in the experimental group | Month 0
  Alkaline phosphatase (ALP) will be measured in units per liter
Alkaline phosphatase in the experimental group | Month 3
  Alkaline phosphatase (ALP) will be measured in units per liter
Alkaline phosphatase in the control group | Month 0
  Alkaline phosphatase (ALP) will be measured in units per liter
Alkaline phosphatase in the control group | Month 3
  Alkaline phosphatase (ALP) will be measured in units per liter
Calcium in the experimental group | Month 0
  Calcium will be measured in mmol/L
Calcium in the experimental group | Month 3
  Calcium will be measured in mmol/L
Calcium in the control group | Month 0
  Calcium will be measured in mmol/L
Calcium in the control group | Month 3
  Calcium will be measured in mmol/L
Creatinine in the experimental group | Month 0
  Calcium will be measured in μmol/L
Creatinine in the experimental group | Month 12
  Calcium will be measured in μmol/L
Creatinine in the control group | Month 0
  Calcium will be measured in μmol/L
Creatinine in the control group | Month 12
  Calcium will be measured in μmol/L
Albumin in the experimental group | Month 0
  Albumin will be measured in g/liter
Albumin in the experimental group | Month 12
  Albumin will be measured in g/liter
Albumin in the control group | Month 0
  Albumin will be measured in g/liter
Albumin in the control group | Month 12
  Albumin will be measured in g/liter
Urea in the experimental group | Month 0
  Urea will be measured in mmol/L
Urea in the experimental group | Month 12
  Urea will be measured in mmol/L
Urea in the control group | Month 0
  Urea will be measured in mmol/L
Urea in the control group | Month 12
  Urea will be measured in mmol/L
Bilirubin in the experimental group | Month 0
  Bilirubin will be measured in µmol/L
Bilirubin in the experimental group | Month 12
  Bilirubin will be measured in µmol/L
Bilirubin in the control group | Month 0
  Bilirubin will be measured in µmol/L
Bilirubin in the control group | Month 12
  Bilirubin will be measured in µmol/L
C-Reactive Protein in the experimental group | Month 0
  C-Reactive Protein will be measured in mg/L
C-Reactive Protein in the experimental group | Month 12
  C-Reactive Protein will be measured in mg/L
C-Reactive Protein in the control group | Month 0
  C-Reactive Protein will be measured in mg/L
C-Reactive Protein in the control group | Month 12
  C-Reactive Protein will be measured in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Cédric LUKAS, Professor, Study Director — Montpellier University Hospital; Jacques MOREL, Professor, Principal Investigator — Montpellier University Hospital; Claire DAIEN, Professor, Principal Investigator — Montpellier University Hospital; Gaël MOUTERDE, Doctor, Principal Investigator — Montpellier University Hospital; Cécile GAUJOUX-VIALA, Professor, Principal Investigator — Nîmes University Hospital; Denis MULLEMAN, Professor, Principal Investigator — Tours University Hospital; Guillermo CARVAJAL, Doctor, Principal Investigator — Tours University Hospital
Locations (3):
- France (3):
  - Nîmes University Hospital, Nîmes, Gard
  - Montpellier University Hospital, Montpellier, Hérault
  - Tours Regional University Hospital (Bretonneau), Tours, Indre-et-Loire

IPD SHARING:
Plan to Share IPD: No